CLINICAL TRIAL: NCT06856278
Title: Clinical Exploratory Study of NKG2D CAR-NK Combined with PD-1 Monoclonal Antibody in the Treatment of Anaplastic Thyroid Cancer (ATC)
Brief Title: Clinical Study of NKG2D CAR-NK Combined with PD-1 Monoclonal Antibody in the Treatment of ATC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR-NK GeT
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-09

CONDITIONS: Anaplastic Throid Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treated with CAR-NK immune cells combined with PD-1 monoclonal antibody. (Experimental)
  Interventions: Drug: NKG2D CAR-NK with PD-1 Antibody

INTERVENTIONS:
Drug: NKG2D CAR-NK with PD-1 Antibody — Treated with CAR-NK immune cells combined with PD-1 monoclonal antibody.

SUMMARY:
The patients with anaplastic thyroid cancer were treated with CAR-NK immune cells combined with PD-1 monoclonal antibody, and the safety and tolerability of the patients were observed and evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years (including boundary values), male or female.
2. Be diagnosed with anaplastic thyroid cancer histopathologically with a measurable lesion≥1cm.
3. Liver and kidney function is good, and can tolerate treatment.
4. Be able to cooperate with the completion of treatment and follow-up work.
5. No other systemic diseases, including other malignancies.

Exclusion Criteria:

1. Need to breastfeed the baby or have fertility needs；
2. Immune system diseases;
3. Diseases of the blood system;
4. Mental system diseases;
5. Interstitial pneumonia, lung disease, etc.;
6. Failure to follow rules of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-22 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | From the start of the trial to day 56 after the first infusion of CAR-NK.
  Safety and tolerability at 28 days after combination therapy, dose limiting toxicity (DLT) and maximum tolerated dose (MTD) were determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No